CLINICAL TRIAL: NCT06381193
Title: Study for the Management of Chronic and Functional Constipation Through the Intake of Probiotics and Prebiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centros de Investigación de Nutrición y Salud (Other)
Collaborators: Nutribiotica (Unknown)
Responsible Party: Principal Investigator, Ismael San Mauro Martin, Principal Investigator, Centros de Investigación de Nutrición y Salud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESTR-01-2022
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Functional Constipation
MeSH Terms: interventions — Probiotics; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental)
  Interventions: Dietary Supplement: Probiotic
- Group B (Experimental)
  Interventions: Dietary Supplement: Prebiotic
- Group C (Experimental)
  Interventions: Dietary Supplement: Probiotic + Prebiotic
- Group D (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — oral, daily
  Arms: Group A
Dietary Supplement: Prebiotic — oral, daily
  Arms: Group B
Dietary Supplement: Probiotic + Prebiotic — oral, daily
  Arms: Group C
Dietary Supplement: Placebo — oral, daily
  Arms: Group D

SUMMARY:
The goal of this clinical trial is to learn if supplementation with prebiotics and/or probiotics can lead to an improvement in symptoms of patients with functional constipation. The main objectives are:

* To evaluate the effect of the dietary supplements on the bowel frequency movements in patients with chronic functional constipation, after 8 weeks.
* To evaluate the stool consistency after 8 weeks (Bristol scale).
* To evaluate the quality of life scale score for patients with Constipation (CVE20 and GSRS scales), after 8 weeks.

Participants are randomized into the following groups:

* Group A: 20 assigned to probiotic + placebo
* Group B: 20 assigned to prebiotic + placebo
* Group C: 20 assigned to probiotic + prebiotic
* Group D: 20 assigned to the placebo + placebo

Participants took 4 units of product per day (2 of each assigned product) for 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between 18-65.
2. BMI 18.5-39.9 kg/m2
3. According to the ROME IV criteria, patients with functional constipation who meet the following conditions for at least the last three months and with symptoms for at least 6 months before diagnosis:

   * The presence of two or more of the following criteria:

     1. Excessive straining at least in 25% of bowel movements.
     2. Hard stools (types 1-2 on the Bristol scale) at least in 25% of stools.
     3. Sensation of incomplete evacuation at least in 25% of the stools.
     4. Sensation of anorectal obstruction or blockage at least in 25% of bowel movements.
     5. Manual maneuvers to facilitate defecation at least in 25% of stools.
     6. Less than three complete spontaneous bowel movements per week.
   * Diarrhea rarely occurs without the use of laxatives.
   * Insufficient criteria for the diagnosis of irritable bowel syndrome.

   Or, according to the ROME IV criteria, patients who suffer from constipation type irritable bowel syndrome defined as a syndrome in which there is abdominal pain with at least two of the following three characteristics:
   * Related to defecation.
   * Associated with change in stool frequency.
   * Associated with a change in stool shape or appearance.
4. Patients who have signed the informed consent.
5. Patients with the ability to understand and carry out the study procedures.
6. Women participating in the study must meet one of these two conditions:

   1. Women without the possibility of becoming pregnant, defined as any woman who has undergone surgical sterilization or is in a postmenopausal state.
   2. Women with the possibility of becoming pregnant who regularly use a highly effective contraceptive method (i.e., hormonal contraception, intrauterine device, condoms, sterilization of the male partner (vasectomy), or complete sexual abstinence) while participating in the study.

Exclusion Criteria:

1. Minors under 18 or over 65 years of age.
2. Patients diagnosed with other chronic diseases ( Parkinson's or other dementias, cerebral palsy, heart attack, tetraplegia, hemiplegia, intellectual disability, multiple sclerosis, amyotrophic lateral sclerosis (ALS), cystic fibrosis, congenital metabolic diseases, eating disorders).
3. With previous surgeries in the gastrointestinal tract.
4. Patients with scheduled surgical interventions during the study.
5. Patient treated with anticoagulants.
6. Patients who have used laxative treatment during the 15 days before the start of the study.
7. Patients who have been treated with antibiotics in the last month.
8. Usual treatment with opioid analgesics.
9. Consumption of supplements with probiotics or prebiotics during the last two weeks before inclusion in the study.
10. Patients diagnosed or with sufficient criteria for the diagnosis of ulcerative colitis, Crohn's disease, presence of intestinal obstruction or malignant disease in the gastrointestinal tract.
11. Participation in another clinical trial with an investigational medication 30 days before the start of the study.
12. Pregnant or breastfeeding women.
13. Patients with hypersensitivity, allergy or intolerance to any of the components of the food supplements in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
1. To evaluate the effect of the dietary supplements on the bowel frequency movements in patients with chronic functional constipation. | 8 weeks

SECONDARY OUTCOMES:
To evaluate the stool consistency (Bristol scale). | 8 weeks
  Type 1-7 (types 3 and 4 indicate a regular transit)
To evaluate the quality of life scale score for patients with constipation (Quality of life questionnaire for patients with constipation, CVE-20) | 8 weeks
To evaluate the quality of life scale score for patients with constipation (Gastrointestinal Symptom Assessment Scale, GSRS scale). | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centros de Investigación en Nutrición y Salud SL. (Clínica CINUSA), Madrid, Spain